CLINICAL TRIAL: NCT05727124
Title: Evaluation of Poul Gjessing Versus T Loops for Orthodontic Maxillary Canine Retraction: A Randomized Clinical Study
Brief Title: Poul Gjessing Versus T Loops for Orthodontic Maxillary Canine Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Saleh Abdullah Mohammed Abdulsalam, BDS(2018) ,Faculty of dentistry, Aden university, Yemen, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 790/2251
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-08

CONDITIONS: Canine Retraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of Poul Gjessing spring for orthodontic maxillary canine retraction (Active Comparator): 20 Orthodontic patient treated by Poul Gjessing spring for canine retraction split mouth.
  Interventions: Device: Poul Gjessing
- Evaluation of T loop for orthodontic maxillary canine retraction (Active Comparator): 20 Orthodontic patient treated by T loop for canine retraction split mouth
  Interventions: Device: T loops

INTERVENTIONS:
Device: Poul Gjessing — maxillary canine retraction
  Arms: Evaluation of Poul Gjessing spring for orthodontic maxillary canine retraction
Device: T loops — T loops
  Arms: Evaluation of T loop for orthodontic maxillary canine retraction

SUMMARY:
Poul Gjessing versus T loops for orthodontic maxillary canine

DETAILED DESCRIPTION:
Split mouth study one side using Poul Gjessing spring and other side using T loops

ELIGIBILITY:
Inclusion Criteria:

* - Class I or II div 1, orthodontic patients, with moderate to severe crowding who are indicated for maxillary first premolar extraction. 2- All permanent teeth are erupted (3rd molars are not included). 3- Good oral and general health. 4- No previous orthodontic treatment.

Exclusion Criteria:

- 1- Orthodontic cases that could be treated with no indication for extraction therapy.

2- Orthodontic cases that are indicate for the extraction of any tooth other than maxillary first premolars. 3- Patients with systemic diseases that might interfere with the of orthodontic tooth movement.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
rate of canine retraction distance | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided